CLINICAL TRIAL: NCT07160192
Title: Monocentric, Non-interventional Study Evaluating the Long-term Outcomes of Percutaneous Endoscopic Caecostomy (PEC) in Patients With Refractory Chronic Constipation
Brief Title: Long-term Evaluation of Percutaneous Endoscopic Caecostomy in Refractory Constipation
Acronym: CONSTICAP 2
Status: Not yet recruiting | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC25_0207
Record Dates: First submitted 2025-06-06; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Constipation; Refractory
Keywords: Caecostomy; Endoscopy; Constipation; GIQLI; Long-term evaluation; SF-36
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Long-term success rate of PEC: Composite outcome: (1) catheter still in place, (2) symptom improvement (GIQLI and KESS), and (3) positive answer to "Would you recommend this technique to someone with the same condition?"

SUMMARY:
This observational monocentric study aims to evaluate the long-term effectiveness and tolerance of percutaneous endoscopic caecostomy (PEC) in patients with chronic refractory constipation. Follow-up data will be collected through phone interviews and standardized quality of life questionnaires.

DETAILED DESCRIPTION:
CONSTICAP 2 is a non-interventional cohort study conducted at CHU de Nantes. Patients who received a PEC between 2010 and 2022 will be contacted by phone at least two years after the procedure. Data will be collected using validated questionnaires (GIQLI, SF-36, etc.) to assess quality of life and treatment durability. The study builds on baseline and short-term data from the CONSTICAPE 1 cohort.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Received PEC at CHU de Nantes
* Affiliated to French social security
* Non-opposition obtained

Exclusion Criteria:

* No PEC placement
* Protected adults or unable to respond
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with refractory constipation treated with PEC at CHU Nantes.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the long-term quality of life of patients | At 2 years of follow-up.
  The assessment of the primary endpoint (long-term quality of life) is based on a composite endpoint (cf. Description Primary Outcomes 1 to 5):
  - Catheter removal: positive if definitive removal without reimplantation at the time of the last update.
Evaluation of the long-term quality of life of patients | At 2 years of follow-up.
  The assessment of the primary endpoint (long-term quality of life) is based on a composite endpointt (cf. Description Primary Outcomes 1 to 5):
  - GIQLI: positive if GIQLI ≥ +10 points vs. baseline.
Evaluation of the long-term quality of life of patients | At 2 years of follow-up.
  The assessment of the primary endpoint (long-term quality of life) is based on a composite endpoint:
  (cf. Description Primary Outcomes 1 to 5):
  - Kess: positive if Kess ≤ -5 points vs. baseline.
Evaluation of the long-term quality of life of patients | At 2 years of follow-up.
  The assessment of the primary endpoint (long-term quality of life) is based on a composite endpoint: (cf. Description Primary Outcomes 1 to 5):
  - Kess: positive if Kess ≤ -5 points vs. baseline.
Evaluation of the long-term quality of life of patients | At 2 years of follow-up.
  The assessment of the primary endpoint (long-term quality of life) is based on a composite endpoint: (cf. Description Primary Outcomes 1 to 5):
  - Rule: composite success = 3/3 positive components.

SECONDARY OUTCOMES:
Assessment of quality of life using the SF-36 scale | Baseline, 1, 3, 6, 9, and 12 months and at 2 years of follow-up.
  Collection of SF36 scores at baseline and at 1, 3, 6, 9, and 12 months (previous Consticape study). Score between 0 and 100 ; the more elevated, better is the outcome.
Assessment of gastrointestinal quality of life using the GIQLI scale (Gastrointestinal Quality of Life Index) | Baseline, 1, 3, 6, 9, and 12 months and at 2 years of follow-up.
  Collection of GIQLI score at baseline and at 1, 3, 6, 9, and 12 months (previous Consticape study).
  Score between 0 and 144; the more elevated, better is the outcome.
Measures constipation severity using the KESS scale ((symptom scoring system for constipation) | Baseline, 1, 3, 6, 9, and 12 months and at 2 years of follow-up.
  Collection of Kess score at baseline and at 1, 3, 6, 9, and 12 months (previous Consticape study).
  Score between 0 and 39; the more elevated, worst is the outcome (severe constipation).
Assesses fecal incontinence using Cleveland scale | Baseline, 1, 3, 6, 9, and 12 months and at 2 years of follow-up.
  Collection of Cleveland score (Cleveland Clinic Fecal Incontinence Score (Jorge-Wexner, CCFIS)) at baseline and at 1, 3, 6, 9, and 12 months (previous Consticape study).
  Score between 0 and 20; the more elevated, worst is the outcome.
Measures neurogenic bowel dysfunction using NBD scale ((Neurogenic Bowel Dysfunction) | Baseline, 1, 3, 6, 9, and 12 months and at 2 years of follow-up.
  For patients with spina bifida and/or spinal cord injuries, Neurogenic Bowel Dysfunction (NBD) scores at 1, 3, 6, 9, and 12 months (previous Consticape study) Score between 0 and 47; the more elevated, worst is the outcome. Validated categories: 0-6 very minor, 7-9 minor, 10-13 moderate, ≥ 14 severe
Complications | Throughout the 12-month follow-up.
  Compilation of possible immediate or delayed complications during follow-up for up to 12 months (previous Consticape study)
Device Tolerance using EVA scale | 15 days, 1, 3, 6, 9, and 12 months and at 2 years
  Visual Analog Scale (VAS) for pain assessment at 15 days, 1, 3, 6, 9, and 12 months (previous Consticape study), collection of any complications and treatments taken by the patient (previous Consticape study and follow-up after at least 2 years) Score between 0 and 10; the more elevated, worst is the outcome. Commonly used categories: ≤ 3.4 mild, 3.5-7.4 moderate, ≥ 7.5 severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared.